CLINICAL TRIAL: NCT04517526
Title: Efficacy and Safety of Platinum-based Chemotherapy + Bevacizumab + Durvalumab, and Salvage SBRT for IV Non-Small Cell Lung Cancer Patients With EGFR Mutations After Failure of First Line Osimertinib：A Multicenter, Prospective, Phase II Clinical Study
Brief Title: Efficacy and Safety of Platinum-based Chemotherapy + Bevacizumab + Durvalumab, and Salvage SBRT for IV Non-Small Cell Lung Cancer Patients With EGFR Mutations After Failure of First Line Osimertinib: A Multicenter, Prospective, Phase II Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBDS-ZL
Record Dates: First submitted 2020-08-16; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Lung Cancer Stage IV，EGFR-mutant，TKI，PD-L1，SBRT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1 (Experimental): pemetrexed (500 mg/m2/d1) + cisplatin/carboplatin (20-25 mg/m2 × 3 days/AUC 5) + bevacizumab (7.5 mg/kg) + durvalumab (10 mg/kg) every 3 weeks for 4 to 6 cycles , followed by bevacizumab and/or durvalumab anti-maintenance therapy until the emergence of treatment-related toxicity or disease progression in the patient, followed by stereotactic radiotherapy to appropriate oligometastatic or oligoprogressive sites
  Interventions: Drug: pemetrexed，cisplatin/carboplatin，bevacizumab，durvalumab，SBRT

INTERVENTIONS:
Drug: pemetrexed，cisplatin/carboplatin，bevacizumab，durvalumab，SBRT — pemetrexed (500 mg/m2/d1) + cisplatin/carboplatin (20-25 mg/m2 × 3 days/AUC 5) + bevacizumab (7.5 mg/kg) + durvalumab (10 mg/kg) every 3 weeks for 4 to 6 cycles after informed consent, followed by bevacizumab and/or durvalumab anti-maintenance therapy until the emergence of what the investigator considers to be treatment-related toxicity or disease progression in the patient, followed by stereotactic radiotherapy to appropriate oligometastatic or oligoprogressive sites.

SUMMARY:
Lung cancer still occupies the highest incidence and mortality rate in the wordwild, and non-small cell lung cancer (NSCLC) accounts for about 80% to 85% of all lung cancers. Currently, immune checkpoint inhibitors targeting PD-1/PD-L1 have become one of the new standard treatments for advanced NSCLC in some molecular subtypes. In the Asian population, EGFR mutations are the most important molecular subtype in lung cancer patients, with an incidence of 39.6% in NSCLC and even more than 50% in adenocarcinoma. EGFR-TKIs are still the first-line treatment for advanced EGFR-mutant NSCLC and can induce a rapid response in this type of NSCLC, but acquired resistance usually occurs between 9 and 16-18 months (three generations of TKI), and the mechanism is complex. Subsequent treatment options are challenging. In contrast, immune checkpoint inhibitors have a specific role in improving the immune status of cancer patients, which may lead to sustained disease control. Clinical studies have shown that the regimen of pemetrexed/platinum-based chemotherapy combined with/PD-L1 inhibitors and bevacizumab has been effective in patients with EGFR-sensitive mutations. Preclinical and clinical studies have shown that EGFR-TKIs can modulate the tumor immune microenvironment and optimize the anti-tumor activity, thus enhancing the benefit of PD-1/PD-L1 inhibitors in patients with NSCLC. In addition, recent studies have shown that stereotactic body radiotherapy (SBRT/SRT) also performs well in the treatment of patients with stage IV NSCLC and can bring survival benefits to patients with advanced disease. We propose to design a prospective, multicenter, phase II clinical study of platinum-containing dual-drug chemotherapy + bevacizumab + SBRT/SRT for EGFR-mutant non-small cell lung cancer with first-line progression of Osimertinib, taking into account the current clinical research status. The Durvalumab regimen consists of 4 to 6 cycles of bevacizumab and/or Durvalumab maintenance therapy until disease progression, with stereotactic radiotherapy to oligoprogression sites, with the ultimate expectation of long-term survival benefit for this group of patients. The primary endpoints are PFS, overall OS, secondary endpoints are treatment-related toxicity, disease control rate, and exploratory endpoints are molecular markers of potential efficacy and toxicity,

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75.
2. Life expectancy exceeding 3 months.
3. Histologic or cytologic pathology confirmed non-small cell lung cancer. However, sputum cytology results alone are not acceptable. The cytology results of tracheal swabbing, tracheal irrigation fluid and needle aspiration are acceptable.
4. The investigator confirms the presence of at least one measurable lesion according to the RECIST 1.1 criteria.
5. According to the International Association for the Study of Lung Cancer and the Joint Committee on American Cancer Classification, 8th Edition, TNM stage of lung cancer with histological or Advanced metastatic or recurrent (stage IV) cytologically proven inoperable and not amenable to radical concurrent radiotherapy or chemotherapy Patients with NSCLC.
6. Eastern Oncology Collaborative Group (ECOG) fitness status score of 0 or 1.
7. Genetic testing suggests EGFR driver gene positivity, which can be accompanied by other driver gene positivity.
8. Tumor progression or inability to tolerate chemotherapeutic response at the most recent evaluation following treatment with Osimertinib.
9. Good hematopoiesis, defined as an absolute neutrophil count ≥1.5 × 109/L, platelet count ≥100 ×109/L，Erythropoietin ≥ 90 g/L [7 days without transfusion or erythropoietin (EPO-dependent).
10. Good liver function, defined as total bilirubin levels ≤ 1.5 times the upper limit of normal (ULN); in patients without hepatic metastases, glutinous rice straw is used as a supplement.
11. Aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN; for patients with documented liver metastases. AST and ALT levels ≤5 times ULN.
12. Good renal function, defined as serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula); less than 2+ urine protein on routine urinalysis, or 24-hour urine protein quantification <1 g.
13. Good coagulation, defined as an International Standardized Ratio (INR) or Prothrombin Time (PT) ≤1.5 times ULN; if the subject is receiving anticoagulant therapy, provided that the PT is within the intended range of use of the anticoagulant.
14. For female subjects of childbearing age, within 3 days prior to receiving the first study drug administration (Week 1, Day 1)A negative urine or serum pregnancy test is performed. If a negative urine pregnancy test cannot be confirmed, a blood pregnancy test may be ordered.
15. High-performance contraception (i.e., methods with a failure rate of less than 1 per cent per year) for both male and female patients if there is a risk of conception.

Exclusion Criteria:

1. NSCLC EGFR driver gene negativity.
2. Pathological examination of a mixture of squamous or small cell lung cancer components.
3. Currently participating in an interventional clinical research treatment or have received another investigational drug within 4 weeks prior to the first administration of the drug.
4. Previous treatment with anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that stimulate or synergistically inhibit another T-cell receptor (e.g., CTLA-4, OX-40, CD137), or radiation therapy in the chest and in metastatic lesions.
5. Systemic systemic therapy with an anti-lung cancer indication with a proprietary Chinese medicine or immunomodulatory drug (including thymidine, interferon, interleukin, except for local use for pleural control) within 2 weeks prior to the first dose, or major surgery within 3 weeks prior to the first dose.
6. Palliative radiotherapy completed within 7 days prior to the first administration of the drug.
7. Presence of clinically active diverticulitis, abdominal abscesses, gastrointestinal obstruction.
8. Have received a transplant of a solid organ or blood system.
9. Presence of clinically uncontrollable pleural effusion/abdominal fluid.
10. Known severe allergic reaction (grade ≥3) to durvalumab, or other immunotherapeutic agents.
11. Active autoimmune disease requiring systemic therapy (e.g., use of disease-modifying drugs, corticosteroids, or immunosuppressants) occurring within 2 years prior to the first dose of the drug. Alternative therapies (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency) are not considered systemic therapy.
12. Diagnosis of immunodeficiency or being on systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days prior to the first administration of the study; physiological doses of glucocorticoids (≤10 mg/day of prednisone or equivalent) are permitted.
13. Have not sufficiently recovered from toxicity and/or complications from any of the interventions prior to initiating treatment (i.e. ≤ grade 1 or at baseline, not including weakness or hair loss).
14. Diagnosis of other malignancies within 5 years prior to the first dose, with exceptions including radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radically resected carcinoma in situ.
15. Symptomatic central nerve metastases. Patients with asymptomatic brain metastases or stable symptoms after treatment of brain metastatic lesions may be enrolled in this study if all of the following criteria are met: measurable lesions outside the central nervous system; absence of midbrain, bridge, cerebellum, medulla oblongata or spinal cord metastases; maintenance of clinical stability for at least 2 weeks; and cessation of hormonal therapy 3 days prior to the first dose of study drug.
16. A history of non-infectious pneumonia requiring glucocorticoid therapy or current interstitial lung disease within 1 year prior to the first administration of the drug.
17. Active infections that require systemic treatment.
18. The known existence of a mental illness or substance abuse condition that may affect compliance with the test requirements.
19. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive).
20. Note: Subjects with hepatitis B who meet the following criteria are also eligible for enrollment: HBV viral load must be <1000 copies/ml (200 IU/ml) prior to first dose and subjects should receive anti-HBV therapy to avoid viral reactivation throughout the duration of study chemotherapy drug therapy. Subjects with anti-HBc (+), HBsAg (-), anti-HB (-) and HBV viral load (-) do not need to receive prophylactic anti-HBV therapy but need to be monitored closely for viral reactivation.
21. Active HCV-infected subjects (HCV antibody-positive and HCV-RNA levels above the lower limit of detection).
22. Live vaccine within 30 days prior to first dose (Cycle 1, Day 1); NOTE: Injectable inactivated viral vaccine against seasonal influenza is allowed up to 30 days prior to first dose; however, live attenuated influenza vaccine for intranasal administration is not allowed.
23. Evidence of a medical history or illness that could interfere with the results of the trial, prevent the subject from participating throughout the study, abnormal values for treatment or laboratory tests, or other circumstances that, in the opinion of the investigator, make enrollment unsuitable.
24. Breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  the time between the start of treatment and the observation of disease progression or the occurrence of death from any cause, in this study there will be two stages of PFS available for analysis. Patients who are still alive at the time of analysis will have the date of their last contact as the cut-off date
Overall survival (OS) | 2 years
  The time from the first day of enrolment to death from any cause, with the date of last contact for patients still alive at the time of analysis as the cut-off date.

SECONDARY OUTCOMES:
overall response rate (ORR) | 2years
  overall remission rate
Duration of response（DOR) | 2years
  duration of remission for all lesions after multi-drug combination therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University shanghai cancer center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided